CLINICAL TRIAL: NCT01321983
Title: Effects of Preoperative Inspiratory Muscle Training (IMT) in Obese Women Undergoing Open Bariatric Surgery: Respiratory Muscle Strength, Lung Volumes and Diaphragmatic Excursion
Brief Title: Effects of Preoperative Inspiratory Muscle Training (IMT) in Obese Women Undergoing Open Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Sao Carlos (Other)
Collaborators: Meridional Hospital (Unknown); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Other Study IDs: 141299/2009-6
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Preoperative Inspiratory Muscular Training; Bariatric Surgery; Chest Physiotherapy; Postoperative Pulmonary Complications; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Inspiratory muscular training - IMT

SUMMARY:
OBJECTIVE: to determine whether preoperative inspiratory muscle training (IMT) is able to attenuate the impact of surgical trauma on the respiratory muscle strength, in the lung volumes and diaphragmatic excursion in obese women undergoing open bariatric surgery.

Therefore, the hypothesis of the present study was that preoperative IMT is able to attenuate the negative effects of surgical trauma on the respiratory muscle strength, in the lung volumes and diaphragmatic excursion, thus reducing the risk of PPC, in obese patients undergoing open bariatric surgery.

DESIGN: Randomized controlled trial. SETTING: Meridional Hospital, Cariacica/ES, Brazil. SUBJECTS: Thirty-two obese women undergoing elective open bariatric surgery were randomly assigned to receive preoperative inspiratory muscle training (IMT group) or usual care (control group).

MAIN MEASURES: Respiratory muscle strength (maximal inspiratory pressure - MIP and maximal expiratory pressure - MEP), lung volumes and diaphragmatic excursion.

ELIGIBILITY:
Inclusion Criteria:

* Female,
* Over 18 years of age,
* No smoking or respiratory disease.

Exclusion Criteria:

* Patients who refused to participate in the steps of the research protocol,
* Patients with a history of prior abdominal surgery,
* Patients who were unable to understand and perform the tests properly
* Patients who refused to sign the Informed Consent Term.

Ages: 18 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Meridional Hospital, Cariacica, Espírito Santo, Brazil

REFERENCES:
- See also: Related Info — http://www.ufscar.br